CLINICAL TRIAL: NCT01240629
Title: A Phase I/II Trial of AN-152 [AEZS-108) in Castration- and Taxane-Resistant Prostate Cancer
Brief Title: Doxorubicin-GnRH Agonist Conjugate AEZS-108 in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4P-09-9; NCI-2009-01418
Record Dates: First submitted 2010-06-30; First posted 2010-11-15 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Prostate Cancer; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — LHRH, lysine(6)-doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive doxorubicin-GnRH agonist conjugate AEZS-108 intravenously (IV) over 2 hours once every 21 days (21 days = 1 cycle). Treatment repeats every 21 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Other: questionnaire administration; Drug: doxorubicin-GnRH agonist conjugate AEZS-108

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative study
Other: questionnaire administration — Correlative study
Drug: doxorubicin-GnRH agonist conjugate AEZS-108 — Given IV
  Other Names: AEZS-108; doxorubicin-LHRH agonist conjugate AEZS-108

SUMMARY:
This is a research study for advanced prostate cancer. An experimental drug called AN-152 (also known as AEZS-108) will be used. The purpose of this study is to test the safety, tolerability and benefits of an experimental drug called AN-152.

The participants tumor will be tested for expression of this receptor (using an old biopsy). If the participants cancer does not have this receptor, participants will not be eligible to participant in this study.

AN-152 (AEZS-108) is administered intravenously (IV) over 2 hours and will be given at the specified dose every 3 weeks. Premedication with dexamethasone 8mg is recommended.

Participants will continue treatment until death, disease progression, unacceptable toxicity, participants refusal, treatment delay >3 weeks, or the completion of 6 cycles. Continuation beyond 6 cycles is left at the discretion of the study doctor.

The study is planned to last 2 years. Up to 55 (up to 18 for the Phase I portion, up to 37 for the Phase II portion).

ELIGIBILITY:
Inclusion

* Histologically or cytologically confirmed prostate cancer
* Measurable disease on computer tomography (CT) scan or evaluable disease with an elevated prostate specific antigen (PSA)
* Documented progression on (a) at least one prior hormone treatment, which must have incorporated luteinizing hormone-releasing hormone (LH- RH)agonist therapy AND (b) at least one chemotherapy regimen, which must have been taxane based
* Progression may be demonstrated by PSA (defined by a 25% increase in the PSA from its most recent treatment nadir, confirmed with a second measurement at least 4 weeks later) or radiologic criteria (defined by radiologic documentation of a new lesion or a >= 20% increase in the sum of the diameters of previously noted measurable lesions)
* Palliative radiation therapy (RT) for metastatic disease is allowed only if =< 25% of total body bone marrow was irradiated and =< 35Gy administered to the pericardial area
* 28 days must have elapsed since completion of RT with bone marrow recovery
* Soft tissue disease irradiated in the prior 2 months may not be designated as measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance score of 0-2
* Adequate bone marrow function, defined by ANC >= 1000/ul, hemoglobin >= 8.0 g/dL and platelet count >= 75,000/ ul
* Adequate renal function, defined by serum creatinine =< 1.5x the upper limit of normal (ULN)
* Adequate hepatic function, defined by bilirubin =< 1.5 mg/dL AND alkaline phosphatase =< 3x ULN for the reference lab (=< 5x ULN for patients with known hepatic metastases and no limit for patients with known bone metastases) AND AST and ALT =< 3x ULN (=< 5x the ULN for patients with known hepatic metastases)
* Must have recovered from acute and late effects of any prior surgery, radiotherapy or other anti-neoplastic therapy
* Patients or their legal representatives must be able to read,understand, and provide informed consent
* Men of childbearing potential must consent to use barrier contraception while on treatment and for 90 days thereafter
* Willingness to discontinue LH-RH analogue therapy and for the duration of the study

Exclusion

* Ongoing use of an LH-RH agonist (or antagonist)
* Patients who agree to stop LH-RH agonist therapy will be eligible but may need to wait until their required washout period is over
* Patients whose washout period is more than 6 weeks will not be eligible
* Duration of washout period varies with the formulation of the LH-RH agonist being used and should be 2 weeks after the next dose would be scheduled. Specifically: a) For patients receiving a monthly formulations of LH-RH agonist, 6 weeks must pass from the last dose before eligibility; b) For patients receiving a 3-month depot formulation of LH-RH agonist, 14 weeks must pass from the last dose before eligibility; c) For patients receiving a 4- month depot formulation of LH-RH agonist, 18 weeks must pass from the last dose before eligibility; d) For patients receiving a 6- month depot formulation of LH-RH agonist, 26 weeks must pass from the last dose before eligibility; e) For patients with an annual LH-RH implant, 2 weeks must pass after removal of the implant before eligibility
* Presence of an active infection or fever within 3 days of the first scheduled protocol treatment
* Presence of parenchymal brain metastases
* Patients with neurological symptoms must have a CT or magnetic resonance imaging (MRI)scan of the brain showing no metastases within 60 days of enrollment
* History of prior malignancy within the past 5 years with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or superficial bladder
* Patients with known hypersensitivity to any of the components of AN-152 including doxorubicin and LH-RH agonists
* Patients who received radiotherapy within 4 weeks of entry
* Patients who received treatment with strontium-89 or samarium-153 are excluded, except prior samarium will be allowed provided it was administered more than 1 year ago and/or the patient has demonstrated the ability to receive cytotoxic chemotherapy without excess of myelosuppression after receiving samarium.
* Patients with a history of unstable or newly diagnosed angina pectoris, documented history of current serious arrhythmia or congestive heart failure or recent myocardial infarction (within 6 months of enrollment)
* Left ventricular ejection fraction (EF) < 50%
* Prior exposure to anthracyclines or anthracenediones including doxorubicin, daunorubicin, and mitoxantrone
* Major surgery within the last 2 weeks
* Receiving concurrent investigational therapy or have received investigational therapy within 30 days of the first scheduled day of protocol treatment (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication)
* Known HIV or hepatitis B or C infection
* Life expectancy < 3 months
* Presence of any other medical condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with interpretation of the results
* Prior treatment with AN-152
* Lack of ability or willingness to give informed consent
* Anticipated non-availability for study visits/procedures

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-11-02 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit defined as non-progression with no dose-limiting toxicity or other toxicity requiring termination of treatment | At 3 months up to 24 months

SECONDARY OUTCOMES:
Time to overall disease progression | Up to 24 months
Response for patients with measurable disease based on the Response Evaluation Criteria in Solid Tumors (RECIST) | At 3 months up to 24 months
To assess the prostate specific antigen (PSA) response rate in patients treated with AN-152 | At 3 months up to 24 months
Time to PSA progression | Up to 24 months
Number of participants with adverse events as a measure of safety and tolerability | At 3 weeks up to 72 weeks
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Pinski, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States